CLINICAL TRIAL: NCT03966937
Title: Effects of Trigger Point Dry Needling In Patient With Patellofemoral Pain Syndrome
Brief Title: Trigger Point Dry Needling In Patient With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahIU Nadia Ishtiaq
Record Dates: First submitted 2019-05-16; First posted 2019-05-29 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Anterior Knee Pain Syndrome; Patellofemoral Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: There will be two treatment groups of participants, One group will receive Dry Needling for releasing trigger points in Quadriceps along with therapeutic exercises whereas other will receive only therapeutic exercises
Who Masked: Participant
Masking Description: This is a single blinded randomized controlled trial in which patients will be randomized into groups by sealed envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): The experimental group will receive dry needling over trigger points of Quadriceps muscles along with therapeutic exercises.
  Interventions: Other: Dry needling
- Control (Active Comparator): The control group will only receive standardized therapeutic exercises for Patellofemoral pain syndrome.
  Interventions: Other: Control

INTERVENTIONS:
Other: Dry needling — Hot Pack will be applied on Quadriceps muscles before session for general relaxation for 7-10 minutes. Stretching of quadriceps femoris muscle with 4 repetitions and 15 second hold per session will be performed. Strengthening exercises of 3 sets of 10 RM with progressive loading per session will be performed.
  Then after wearing gloves and appropriate personal protective measures, a thin filiform needle will be inserted which will penetrate into the skin and stimulate underlying myofascial trigger points.
  Arms: Dry needling
Other: Control — Hot Pack will be applied on Quadriceps muscles before session for general relaxation for 7-10 minutes. Stretching of quadriceps femoris muscle with 4 repetitions and 15 second hold per session will be performed. Strengthening exercises of 3 sets of 10 RM with progressive loading per session will be performed.
  Arms: Control

SUMMARY:
This study intends to determine the effects of trigger point dry needling in patients with Patellofemoral pain Syndrome.

DETAILED DESCRIPTION:
This is a single blinded randomized controlled trial, will be conducted at District Head Quarter (DHQ) hospital Taunsa Sharif.

Dry needling is a technique used to release myofascial trigger points. this study is planned to determine the effects of dry needling on quadriceps muscle in patients with Patellofemoral pain syndrome. The sample size was calculated to be n=92 through Open Epi tool version 3, with 95 % confidence interval (CI), and power 80%,

After the completion of therapeutic protocols, the participants will be assessed with the help of Numeric Pain Rating Scale (NPRS), Algometer and Anterior Knee Pain scale along with knee Range of Motion(ROM)

ELIGIBILITY:
Inclusion Criteria:

* Males and females with age limit 20 to 40 years,
* Active knee extension/90-90 test positive for Screening (With AKE range less than 160 degrees),
* No known history of hip joint or knee joint disease,
* No history of recent hamstring strain.

Exclusion Criteria:

* Patient with meniscal tears, patellar tendinopathy, and ligamentous injuries.
* Patient with knee osteoarthritis
* Patient with lumbosacral nerve root or peripheral nerve involvement

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Numeric Pain Rating Scale (NPRS) | Post 1st week
  Numeric Pain Rating Scale (NPRS) is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Algometer | Baseline
  Pressure threshold is the minimal pressure (force) which induces pain. The digital algometer is a force gauge with a rubber disc of 1 cm2 surface. It will be placed over trigger point in muscle and pressure pain sensitivity would be measured.
Algometer | Post 1st week
  Pressure threshold is the minimal pressure (force) which induces pain. The digital algometer is a force gauge with a rubber disc of 1 cm2 surface. It will be placed over trigger point in muscle and pressure pain sensitivity would be measured.
Anterior Knee Pain Scale (AKPS) | Baseline
  The Anterior Knee Pain Scale (AKPS) - sometimes called the Kujala Scale is a 13-item knee-specific self-report questionnaire. It documents response to six activities (walking, running, jumping, climbing stairs, squatting, and sitting for prolonged periods with knees bent), as well as symptoms such as limp.
  The maximum score is 100 that indicate good results, if score is 70 then it is moderate, lower scores like 50 or below 50 indicates severity of the disease.
Anterior Knee Pain Scale (AKPS) | Post 1st week
  The Anterior Knee Pain Scale (AKPS) - sometimes called the Kujala Scale is a 13-item knee-specific self-report questionnaire. It documents response to six activities (walking, running, jumping, climbing stairs, squatting, and sitting for prolonged periods with knees bent), as well as symptoms such as limp.
  The maximum score is 100 that indicate good results, if score is 70 then it is moderate, lower scores like 50 or below 50 indicates severity of the disease.
Knee Range of Motion (ROM) | Baseline
  To assess Knee range of motion (ROM), Goniometer will be use to measure knee range of motion in flexion & extension. Participants will be seated upright and asked to actively move their knee in each direction.
Knee Range of Motion (ROM) | Post 1st week
  To assess Knee range of motion (ROM), Goniometer will be use to measure knee range of motion in flexion & extension. Participants will be seated upright and asked to actively move their knee in each direction.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- District Health Quarter Taunsa, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boling M, Padua D, Marshall S, Guskiewicz K, Pyne S, Beutler A. Gender differences in the incidence and prevalence of patellofemoral pain syndrome. Scand J Med Sci Sports. 2010 Oct;20(5):725-30. doi: 10.1111/j.1600-0838.2009.00996.x. PMID 19765240
- [Background] Collado H, Fredericson M. Patellofemoral pain syndrome. Clin Sports Med. 2010 Jul;29(3):379-98. doi: 10.1016/j.csm.2010.03.012. PMID 20610028
- [Background] Saltychev M, Dutton RA, Laimi K, Beaupre GS, Virolainen P, Fredericson M. Effectiveness of conservative treatment for patellofemoral pain syndrome: A systematic review and meta-analysis. J Rehabil Med. 2018 May 8;50(5):393-401. doi: 10.2340/16501977-2295. PMID 29392329
- [Background] Starkweather A. The Evidence on Dry Needling for Pain Management.Topics in Pain Management. 2018 Nov 1;34(4):1-9
- [Background] Sutlive TG, Golden A, King K, Morris WB, Morrison JE, Moore JH, Koppenhaver S. SHORT-TERM EFFECTS OF TRIGGER POINT DRY NEEDLING ON PAIN AND DISABILITY IN SUBJECTS WITH PATELLOFEMORAL PAIN SYNDROME. Int J Sports Phys Ther. 2018 Jun;13(3):462-473. PMID 30038832